CLINICAL TRIAL: NCT00698295
Title: Study of the Relationship Between EEG and Clinical Changes in Drug-Naive or Drug-Free Patients With Schizophrenia After Atypical Antipsychotic Treatment Based on Linear and Non-Linear EEG Analysis
Brief Title: Linear and Non-linear Analysis of EEG Changes in Schizophrenia After Atypical Antipsychotics Medication
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Yong-in Mental Hospital (Unknown)
Responsible Party: Yong Min Ahn/Associate Professor, Seoul National University Hospital
Other Study IDs: 09-2003-009-0
Record Dates: First submitted 2008-06-15; First posted 2008-06-17 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; atypical antipsychotics; EEG
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — routine lab for changes in medical condition
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate clinical meaning of EEG changes in antipsychotic-treated patients with schizophrenia.

DETAILED DESCRIPTION:
Electroencephalographic (EEG) changes are abundant in patients receiving antipsychotic treatment. However, studies on the meaning of these changes are rare. The results of traditional analyses based on linear methodologies were inconsistent and hard to interpret. Therefore, non-linear analyses of EEG may provide additional information in evaluating antipsychotic-induced changes in EEG.

In this study, we hypothesized that linear and non-linear EEG changes in patients with schizophrenia may be valuable in predicting treatment outcome. We also hypothesized that the assessment of other psychotic symptoms and side effects of antipsychotics may provide additional information in interpreting the results of EEG analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 15-65 years of age.
* Patients must have a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
* Patients who are drug-naive or drug-free for more than 4 weeks.
* Patients who are scheduled to receive atypical antipsychotics.
* Each patient must provide written informed consent after full explanation of study protocol, and authorized legal guardian must understand the nature of the study and must also give assent to study participation.
* Subjects who are fluent in Korean.

Exclusion Criteria:

* DSM-IV substance (except nicotine or caffeine) dependence within the past 1 year.
* Mental retardation (IQ < 70).
* Neurological disorders including epilepsy, stroke, or severe head trauma.
* Clinically significant laboratory abnormalities, on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, urinalysis and EKG.
* Treatment with an injectable depot neuroleptic within less than three dosing interval between the last depot neuroleptic injections and baseline.
* History of electroconvulsive therapy or transcranial magnetic stimulation within the past 3 months.
* Subjects who are not fluent in Korean.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with schizophrenia receiving antipsychotic treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2004-09; Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sik Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Yong-in Mental Hospital, Yongin City, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Higashima M, Takeda T, Kikuchi M, Nagasawa T, Koshino Y. Functional connectivity between hemispheres and schizophrenic symptoms: a longitudinal study of interhemispheric EEG coherence in patients with acute exacerbations of schizophrenia. Clin EEG Neurosci. 2006 Jan;37(1):10-5. doi: 10.1177/155005940603700104. PMID 16475479
- [Background] Harris A, Melkonian D, Williams L, Gordon E. Dynamic spectral analysis findings in first episode and chronic schizophrenia. Int J Neurosci. 2006 Mar;116(3):223-46. doi: 10.1080/00207450500402977. PMID 16484051
- [Background] Breakspear M. The nonlinear theory of schizophrenia. Aust N Z J Psychiatry. 2006 Jan;40(1):20-35. doi: 10.1080/j.1440-1614.2006.01737.x. PMID 16403034
- [Background] Wichniak A, Szafranski T, Wierzbicka A, Waliniowska E, Jernajczyk W. Electroencephalogram slowing, sleepiness and treatment response in patients with schizophrenia during olanzapine treatment. J Psychopharmacol. 2006 Jan;20(1):80-5. doi: 10.1177/0269881105056657. Epub 2005 Oct 4. PMID 16204327
- [Background] Chung SJ, Jeong SH, Ahn YM, Kang UG, Koo YJ, Ha JH, Lee SG, Kim YS. A retrospective study of clozapine and electroencephalographic abnormalities in schizophrenic patients. Prog Neuropsychopharmacol Biol Psychiatry. 2002 Jan;26(1):139-44. doi: 10.1016/s0278-5846(01)00238-x. PMID 11853104
- [Background] Kang UG, Par KT, Ahn YM, Koo YJ, Yoon SC, Yi SH, Kim YS. Non-linear dynamic analysis of clozapine-induced electroencephalographic changes in schizophrenic patients--a preliminary study. Prog Neuropsychopharmacol Biol Psychiatry. 2001 Aug;25(6):1229-39. doi: 10.1016/s0278-5846(01)00183-x. PMID 11474842
- See also: Click here for brief explanation of the relationship between schizophrenia and EEG. — http://www.acnp.org/g4/GN401000119/CH117.html
- See also: Click here for concise explanation of the meaning of EEG test in schizophrenia. — http://www.schizophrenia.com/sznews/archives/002206.html